CLINICAL TRIAL: NCT05029349
Title: Exploration of the VOLATOLOM in the Stable Severe COPD (Chronic Obstructive Pulmonary Disease)
Acronym: VOC-BPCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hopital Foch (Other)
Collaborators: Air Liquide SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020_0003
Record Dates: First submitted 2021-07-07; First posted 2021-08-31 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Chronic Obstructive Pulmonary Disease Severe
Keywords: Chronic Obstructive Pulmonary Disease (COPD); Volatile Organic Compounds (VOC); Severe; Stable
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VOC analysis (Other): VOC analysis in exhaled air in patients hospitalised for stable severe COPD
  Interventions: Device: VOC analysis

INTERVENTIONS:
Device: VOC analysis — VOC analysis in exhaled air with e-noses and mass spectrometry.

SUMMARY:
This is a prospective interventional study to determine whether the profile of volatile organic compounds (VOCs) present in exhaled air (VOLATOLOM) is reproducible in stable severe COPD (Chronic Obstructive Pulmonary Disease) patients.

DETAILED DESCRIPTION:
After being informed about the study, all patients giving written informed consent and meeting the eligibility criteria will undergo 4 visits spaced 4 to 6 weeks apart.

The first visit V1 will be about 45 minutes duration. The others ones (V2 to V4) will be about 30 minutes duration.

All sessions will be carried out in the Pneumology Department of the Foch Hospital, volatolomics platform (Exhalomics®).

Exhalation collection will be performed at each visit in order to perform the volatolom analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Severe COPD (FEV ≤ 50% of theoretical values)

   * stable for at least two months,
   * treated for at least one year with one (or more successively) combination of at least two inhaled drugs: either a Long-Acting Beta2-Adrenergic bronchodilator (LABA) combined with a corticosteroid (CSI), or a LABA combined with a long-acting anti-cholinergic bronchodilator (LAMA), or a triple combination LABA/LAMA/CSI;
2. History of at least one severe COPD exacerbation (treated with antibiotics and / or oral corticosteroid therapy) in the two years preceding the study;
3. Ex-smokers (at least 6 months of withdrawal) or active daily smokers of more than 10 pack-years
4. Severe dyspnea at baseline (mMRC stage ≥ 2)
5. Aged 40-85 years inclusive
6. Fluency in French
7. A signed and dated written informed consent is obtained prior to participation
8. Affiliated to a health insurance plan

Exclusion Criteria:

1. Severe exacerbation in the 4 months preceding the study
2. Chronic inflammatory disease (rheumatic, etc.) treated with long-term systemic corticosteroid therapy,
3. Long-term oxygen therapy (exclusive ambulatory oxygen therapy is not a non-inclusion criterion)
4. Unstable cardiovascular pathology (right or left heart failure, coronary artery disease);
5. Cancer
6. Pregnant women;
7. Deprived of liberty or under guardianship.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-10-13 (Actual); Primary Completion 2023-06-13 (Estimated); Study Completion 2023-06-13 (Estimated)

PRIMARY OUTCOMES:
Volatolom measurements by mass spectrometry | 4 months
  Analysis of the volatolom by mass spectrometry for stable severe COPD patients during four successive visits, 4 to 6 weeks apart.
Volatolom measurements by electronic-noses | 4 months
  Analysis of the volatolom by electronic noses for stable severe COPD patients during four successive visits, 4 to 6 weeks apart.

SECONDARY OUTCOMES:
Differences in the profiles of VOCs in the exhaled air according to the smoking habits | 4 months
  Analyze the differences in the exhaled VOCs prints generated by the eNoses and mass spectrometry data processed with the ptairMS R package (https://github.com/camilleroquencourt/ptairMS) according to smoking habits (ex-smokers versus active smokers),
Differences in the profiles of VOCs in the exhaled air according to the background therapy | 4 months
  Analyze the differences in the exhaled VOCs prints generated by the eNoses and mass spectrometry data processed with the ptairMS R package (https://github.com/camilleroquencourt/ptairMS) according to the backgrounf therapy (with or without antibiotic/ oral corticosteroid therapy...)
Compare VOCs profiles in the exhaled air to those of patients with exhacerbated COPD (VOC-BPCO-Exa study sponsored by Hopital Foch) | 4 months
  Comparison of the exhaled VOCs prints generated by the eNoses and mass spectrometry data processed with the ptairMS R package (https://github.com/camilleroquencourt/ptairMS) determined from severe COPD patients at stable state included in the study versus VOCs profiles of patients with exhacerbated COPD (VOC-BPCO-Exa study sponsored by Hopital Foch)
Compare VOCs profiles in the exhaled air to those of healthy subjects smokers or non-smokers (VOLATOPNEE study sponsored by Hopital Foch) | 4 months
  Comparison of the exhaled VOCs prints generated by the eNoses and mass spectrometry data processed with the ptairMS R package (https://github.com/camilleroquencourt/ptairMS) determined from severe COPD patients at stable state included in the study versus VOCs profiles of healthy subjects smokers or non-smokers (VOLATOPNEE study sponsored by Hopital Foch)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Devillier, MD PhD, Principal Investigator — Hopital Foch
Locations (1):
- Foch hospital, Suresnes, France